CLINICAL TRIAL: NCT07339904
Title: ProLARS Trial: Prospective Longitudinal Follow-up of Low Anterior Resection Syndrome (LARS) and COREFO Score After Rectum Surgery in Patients Undergoing Upfront Surgery or Different Neo-adjuvant Treatment Regimens
Acronym: ProLARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Niels Komen, MD, PhD, Head of the Abdominal Surgery Department, Principal Investigator, Clinical Professor, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 6510
Record Dates: First submitted 2025-04-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Rectal Adenocarcinoma; LARS - Low Anterior Resection Syndrome; Rectal Resection; Low Anterior Resection; Total Mesorectal Excision
Keywords: LARS; Rectal resection; Total mesorectal excision; Low anterior resection; Rectal carcinoma
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Patients receive online questionnaires regarding LARS- and COREFO-scores
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront surgery (Other): Patients who undergo rectal resection without neo-adjuvant therapy
  Interventions: Other: Questionnaire
- Neo-adjuvant therapy (Other): Patients who receive neo-adjuvant therapy before undergoing rectal surgery
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Online questionnaire regarding LARS- and COREFO-scores, quality of defecation process, incapacity for work and initiation of treatment for potential LARS at different moments in time

SUMMARY:
OBJECTIVE Low anterior resection syndrome (LARS) is a term for functional bowel complaints occurring after low anterior resection. Symptoms can range from faecal incontinence and frequent loose stools to urgency and incomplete emptying with great impact on quality of life. Little is known about the longitudinal evolution of LARS and the impact of different schedules of neoadjuvant chemoradiotherapy combined with surgery.

The investigators aim to investigate the incidence and evolution of functional bowel complaints in function of different neoadjuvant treatment regimens, type of surgery and adjuvant therapy in patients who undergo surgery for rectal cancer. The investigators focus on following objectives: evolution of LARS- and COREFO-scores per treatment regimen and their impact on work incapacity; identification of possible risk factors potentially related to functional outcome; monitoring and treatment of LARS.

METHODS This will be a multicentre prospective interventional study. The study population will consist of adult patients with rectal cancer, regardless of any neo-adjuvant therapy. Patients will be included for 5 years with a 2 year postoperative follow-up. Interim analysis will be made after 2 years of inclusion. Patients with intellectual disability or clinical colon obstruction are excluded. Automated online questionnaires including LARS and COREFO scores, incapacity for work and defecation quality will be sent at different time points (figure 1) using REDCap.

RESULTS and CONCLUSIONS Longitudinal change of LARS- and COREFO-scores will be visually summarized. Patient, disease or procedure specific risk factors will be assessed as well.

LARS is proven to be the principal postoperative problem after rectal surgery. If the investigators can predict the severity of LARS (minor or major LARS), this can be extremely helpful in deciding whether to perform a sphincter-sparing resection or a rectal amputation instead. Furthermore, the investigators want to offer perspective to patients who are susceptible to a disturbed postoperative bowel function.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Diagnosis of rectal cancer, discussed at the multidisciplinary consultation, with the intention to perform a sphincter preserving total mesorectal excision (TME) or partial mesorectal excision (PME), regardless of the need of neoadjuvant treatment.

Exclusion Criteria:

* History of inflammatory bowel disease (Crohn's disease, ulcerative colitis) due to often persistent bowel complaints and therefore distorted baseline and follow-up data.
* Dementia or intellectual disability.
* Patients who are obstructive and in need a decompressive stoma or rectal stenting due to the lack of baseline data as they are often admitted to the hospital in an urgent setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
The evolution of the COREFO-score (Colorectal Functional Outcome questionnaire) at 2 years after rectal surgery compared to baseline (absolute difference) will be examined | 2 years from when rectal resection or stoma reversal was performed
  27 questions on 5-point Likert scale Higher score = worse bowel function

SECONDARY OUTCOMES:
Evolution of LARS-score (low anterior resection syndrome) at 2 years after rectal surgery compared to baseline (absolute difference) | 2 years from when rectal resection or stoma reversal was performed
  0-20 = no LARS 21-29 = minor LARS 30-42 = major LARS
The evolution of the LARS-score (low anterior resection syndrome) at 2 years after rectal surgery compared to baseline (relative difference) will be examined. | 2 years from when rectal resection or stoma reversal was performed
  0-20 = no LARS 21-29 = minor LARS 30-42 = major LARS
The evolution of the COREFO-score (Colorectal Functional Outcome questionnaire) at 2 years after rectal surgery compared to baseline (relative difference) will be examined | 2 years from when rectal resection or stoma reversal was performed
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100)
The evolution of the LARS-score (low anterior resection syndrome) in the absence of baseline data will be examined as well (absolute difference), comparing 2-year outcome to earliest results. | 2 years from when rectal resection or stoma reversal was performed
  0-20 no LARS 21-29 minor LARS 30-42 major LARS (min 0 - max 42)
The evolution of the LARS-score (low anterior resection syndrome) in the absence of baseline data will be examined as well (relative difference), comparing 2-year outcome to earliest results. | 2 years from when rectal resection or stoma reversal was performed
  0-20 no LARS 21-29 minor LARS 30-42 major LARS (min 0 - max 42)
The evolution of the COREFO-score (Colorectal Functional Outcome questionnaire) in the absence of baseline data will be examined as well (absolute difference), comparing 2-year outcome to earliest results. | 2 years from when rectal resection or stoma reversal was performed
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100)
The evolution of the COREFO-score (Colorectal Functional Outcome questionnaire) in the absence of baseline data will be examined as well (relative difference), comparing 2-year outcome to earliest results. | 2 years from when rectal resection or stoma reversal was performed
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100)
LARS-score (low anterior resection syndrome) score at diagnosis | At diagnosis = baseline
  0-20 no LARS 21-29 minor LARS 30-42 major LARS (min 0 - max 42) LARS = low anterior resection syndrome Using a questionnaire Unit = mean score (0-42)
COREFO-score at diagnosis (Colorectal Functional Outcome questionnaire) | At diagnosis = baseline
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100) COREFO = Colorectal Functional Outcome questionnaire Using a questionnaire Unit = mean score (0-100)
LARS-score (low anterior resection syndrome) after neo-adjuvant therapy | After neo-adjuvant therapy (up to 6 months from baseline)
  0-20 no LARS 21-29 minor LARS 30-42 major LARS (min 0 - max 42) LARS = low anterior resection syndrome Using a questionnaire Unit = mean score (0-42)
COREFO-score after neo-adjuvant therapy (Colorectal Functional Outcome questionnaire) | After neo-adjuvant therapy (up to 6 months from baseline)
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100) COREFO = Colorectal Functional Outcome questionnaire Using a questionnaire Unit = mean score (0-100)
LARS-score (low anterior resection syndrome) shortly prior to surgery when there is a delay of 4 or more weeks after finishing neoadjuvant therapy | 2 days prior to surgery
  0-20 no LARS 21-29 minor LARS 30-42 major LARS (min 0 - max 42) LARS = low anterior resection syndrome Using a questionnaire Unit = mean score (0-42)
COREFO-score (Colorectal Functional Outcome questionnaire) shortly prior to surgery when there is a delay of 4 or more weeks after finishing neoadjuvant therapy | 2 days prior to surgery
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100) COREFO = Colorectal Functional Outcome questionnaire Using a questionnaire Unit = mean score (0-100)
LARS-scores (low anterior resection syndrome) postoperatively after 1 month, 3 months, 6 months, 1 year and 2 years | Postoperatively after 1 month, 3 months, 6 months, 1 year and 2 years
  0-20 no LARS 21-29 minor LARS 30-42 major LARS (min 0 - max 42) LARS = low anterior resection syndrome Using a questionnaire Unit = mean score (0-42)
COREFO-scores (Colorectal Functional Outcome questionnaire) postoperatively after 1 month, 3 months, 6 months, 1 year and 2 years | Postoperatively after 1 month, 3 months, 6 months, 1 year and 2 years
  27 questions on 5-point Likert scale Higher score = worse bowel function (min 0 - max 100) COREFO = Colorectal Functional Outcome questionnaire Using a questionnaire Unit = mean score (0-100)
Evolution of quality of defecation process | 2 years after rectal resection or stoma reversal
  Visual analogue scale 0-10 0 = worst defecation ever 10 = best defecation ever
Incapacity for work | At diagnose (baseline), 2 days after radiotherapy, 1 week after chemotherapy and 1 month after rectal resection
  Time (days) between date of start work incapacity and date back to work (if not yet retired)
Initiation of treatment for potential LARS (low anterior resection syndrome) during follow-up | Up to 2 years after rectal resection
  Yes/no:
  * Dietary measures
  * Medication (probiotics, antidiarrheals, ...)
  * Pelvic floor physiotherapy
  * Transanal irrigation, rectal irrigation, enema
  * Neuromodulation (neurostimulator)
  * Other
  Calculating proportion of patients who received treatment for LARS

OTHER OUTCOMES:
Gender | Baseline
  Male, female, other
Year of birth | Baseline
  Year of birth
Age | Baseline to date of surgery
  Age at diagnosis and at surgery
Hospital admission data | After rectal resection
  Length of stay in days (date of admission for rectal resection until date of dismission)
Medical history | Baseline
  Smoking, diabetes mellitus, abdominal, cardiac, pulmonary (yes/no)
Anthropometry | Baseline
  Body mass index (kg/m²)
Tumor location | After restaging prior to surgery
  Distance in cm from recto-anal angle, based on MRI
Presence of lateral lymph nodes | After restaging prior to surgery
  Presence of lateral lymph nodes (yes/no)
cTNM | After restaging prior to surgery
  Clinical TNM classification of tumor:
  * T: tumor size
  * N: nodal involvement
  * M: metastasis
Percentage of rectal circumference involved | After restaging prior to surgery
  Percentage of rectal circumference involved: on imaging (CT/MRI), coloscopy or ultrasound-endoscopy
Circumferential resection margin | After restaging prior to surgery
  Circumferential resection margin (CRM; on MRI; measured from gland; in mm)
Neoadjuvant therapy | From baseline to surgery
  The eventual use of neoadjuvant therapy: radiotherapy (RT), chemotherapy (CT) (yes/no)
Radiotherapy dose | From baseline to surgery
  Radiotherapy dose (Gy)
Chemotherapy type and frequency | From baseline to surgery
  Certain type of chemotherapy, used for certain amount of cycles
Surgical approach | At surgery
  Surgical approach:
  * Open
  * Laparoscopy
  * Robot
  * Transanal (TaTME)
Configuration of anastomosis | At surgery
  Configuration of colorectal/coloanal anastomosis:
  * End-to-End
  * Side-to-End
  * End-to-Side
  * Side-to-Side
Manual or stapled anastomosis | At surgery
  Manual or stapled anastomosis
Conversion | At surgery
  Conversion during surgery:
  * Robot to laparoscopy (yes/no)
  * Laparoscopy to open (yes/no)
Diverting ileostomy | At surgery
  Use of a diverting ileostomy (yes/no)
Baseline CEA | At baseline
  Baseline CEA: Carcinoembryonic antigen (µg/L)
Histology type | After surgery
  Histology type of tumor (adenocarcinoma, squamous cell carcinoma, neuro-endocrine tumor etc.)
Tumor differentiation | After surgery
  Well differentiated Moderately differentiated poorly differentiated
Tumor perforation | After surgery
  Tumor perforation on histology (yes/no)
Radical resection | After surgery
  Radical resection: R0, R1, R2
pTNM | After surgery
  Pathological TNM classification of tumor
  * T: tumor size
  * N: nodal involvement
  * M: metastasis
Disease free interval | Up to 2 years after rectal resection
  Disease free interval: the period of time between the primary treatment of a malignancy and the first sign of tumor recurrence (in months)
Type of complication | After rectal resection during admission
  Type of complication:
  * Urinary tract infection
  * Pulmonary complications
  * Surgical site infection
  * Intra-abdominal collections/abscess
  * Eventration/evisceration
  * Ileus
  * Small bowel obstruction
  * Anastomotic leakage
  * Deep venous thrombosis
  * Postoperative bleeding
  * Acute renal failure
  * High output ileostomy
  * Other stoma related complications
  * Other (yes/no)
Early complications | Between surgery and 30 days after surgery
  Early complications: before 30 days after surgery
Late complications | From 30 days after surgery up to 2 years after surgery
  Late complications: more than 30 days after surgery
Anastomotic leakage | Up to 3 months after surgery
  Definition of anastomotic leakage:
  * Clinically manifest insufficiency of the anastomosis leading to a clinical state requiring treatment, diagnosed in accordance with surgical practice guidelines by a senior surgeon (no additional or systematic routine iconography nor colonoscopy)
  * Radiological evidence of anastomotic leakage if the patient is clinically symptomatic. Fistulas communicating with the anastomosis on CT scan are classified as AL together with presacral abscesses if extravasation of the colonic contrast is visible on radiological imaging (ref. SAFE 2019 Clinical Investigation Plan)
  (yes/no)
Clavien-Dindo classification | After admission for rectal resection
  Clavien-Dindo classification (grade 0, I, II, IIIa, IIIb, IVa, IVb, V):
  Grade I:
  Minor deviation from normal course; no drugs or interventions needed (only supportive care).
  Grade II:
  Requires pharmacological treatment (e.g. antibiotics, blood transfusion, TPN).
  Grade III:
  Requires surgical, endoscopic, or radiological intervention IIIa: without general anesthesia IIIb: with general anesthesia
  Grade IV:
  Life-threatening complication requiring ICU care IVa: single-organ dysfunction IVb: multi-organ dysfunction
  Grade V:
  Death
CCI-score | After admission for rectal resection
  CCI-score: comprehensive complication index (score from 0-100 calculated with online calculator: https://www.cci-calculator.com/cci-calculator)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Komen, MD PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided